CLINICAL TRIAL: NCT04593303
Title: Validity of Internal Iliac Artery Ligation With Cervico Isthmic Compression Suture During Conservative Management of Placenta Accreta Spectrum
Brief Title: Internal Iliac Artery Ligation During Management of Placenta Accreta Spectrum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University Hospital (Other)
Responsible Party: Principal Investigator, Mohamed Taman, Consultant, Mansoura University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MS.20.09.1255
Record Dates: First submitted 2020-10-12; First posted 2020-10-19 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Placenta Accreta
Keywords: placenta accrete spectrum
MeSH Terms: conditions — Placenta Accreta

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internal iliac artery group (Active Comparator): Bilateral internal Iliac artery ligation will be done followed by urinary bladder dissection then bilateral uterine artery ligation then manual removal of the placenta then cervico isthmic compression suture. (holding the upper border of the cervix by 4 Allis's forceps then suturing the cervix with the anterior uterine wall using continuous suture), Nelaton catheter18 gauge or Hegar's dilator will be inserted inside cervical canal during Cervico isthmic tamponed suture to ensure patency of cervical canal. .
  Interventions: Procedure: Internal iliac artery ligation with cervicoisthmic compression suture
- No internal iliac artery group (Other): Bladder dissection then bilateral uterine artery ligation then cervico isthmic suture without internal iliac artery ligation
  Interventions: Procedure: Cervicoisthmic compression suture without Internal iliac artery ligation

INTERVENTIONS:
Procedure: Internal iliac artery ligation with cervicoisthmic compression suture — Retroperitoneal approach will be performed to ligate both internal iliac arteries before bladder dissection followed by cervicoisthmic compression suture application at placental bed
  Arms: Internal iliac artery group
Procedure: Cervicoisthmic compression suture without Internal iliac artery ligation — Bladder dissection followed by cervicoisthmic compression suture application at placental bed without Internal iliac artery ligation
  Arms: No internal iliac artery group

SUMMARY:
Vessels ligation have been used as a part of conservative management in treatment of placenta accrete spectrum to decrease blood loss as uterine artery ligation and internal iliac artery ligation. Surgical ligation of the anterior divisions of the internal iliac artery is practiced by many tertiary care centers during management of women with PAS disorders. However there is no recommendation toward the routine use of internal iliac artery ligation before bladder dissection during conservative management of (placenta accrete spectrum). The retroperitoneal space will be dissected and bifurcation of common iliac vessels will be identified, After identifying the ureter, the internal iliac artery will be dissected on both sides away from surrounding tissues and from adjacent iliac vein. The anterior branch of each internal iliac artery will be then prophylactically ligated using suture ligation approximately 2-3 cm distal to common iliac artery bifurcation in order to avoid ligation of the posterior division. Principal investigators will conduct a study to evaluate the efficacy of internal iliac artery ligation before bladder dissection during conservative management using cervico isthmic compression suture in cases of Placenta accrete spectrum.

DETAILED DESCRIPTION:
Surgical technique for all participants will be (Cervico isthmic compression suture)

Steps:

* Abdominal wall Incision will be done either in the midline or transverse suprapubic incision.
* Opening the abdominal wall in layers.
* Uterine incision will be done at the upper border of the placenta determined at laparotomy by naked eye.
* Delivery of the baby. Then the placenta will be left in place till doing devascularisation and bladder dissection
* Participants then will be, divided into two groups Participants in internal iliac group will undergo internal iliac artery ligation before bladder dissection Participants in no internal iliac artery group will undergo bladder dissection immediately without internal iliac artery ligation

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant female age between 18_35 years.
2. History of ' 3 caesarean deliveries or less .
3. Pregnant female diagnosed to have none complicated medical disorders e.g. Uncontrolled hypertension, Uncontrolled preeclampsia, Uncontrolled Diabetes mellitus .
4. If ≥2 of the following criteria present by trans abdominal ultrasound and color Doppler examination:

   a-Loss of clear zone c-Placental lacunae. e-Placental bulge. g-Utero-vesical. hyper vascularity. i-Bridging vessels. b-Myometrial thinning. d-Bladder wall interruption. f-Focal exophytic mass. h-Subplacental.hyper vascularity. j-Lacunae feeder vessels.
5. Placenta increta or percreta according to FIGO classification (2019)including:

1. Grade II(FIGO 2019 ) 8:Abnormally invasive placenta (Increta)

Clinical criteria):

At laparotomy Abnormal macroscopic findings over the placental bed: bluish/purple coloring, distension (placental "bulge").

Significant amounts of hyper vascularity (dense tangled bed of vessels or multiple vessels running parallel craniocaudally in the uterine serosa).

No placental tissue seen to be invading through the uterine serosa. Gentle cord traction results in the uterus being pulled inwards without separation of the placenta (so-called the dimple sign).

Histologic criteria:

Hysterectomy specimen or partial myometrial resection of the increta area shows placental villi within the muscular fibers and sometimes in the lumen of the deep uterine vasculature (radial or arcuate arteries),if failed conservative therapy.

2. Grade III(FIGO 2019)8: Abnormally invasive placenta (Percreta) Grade 3a: Limited to the uterine serosa Clinical criteria At laparotomy Abnormal macroscopic findings on uterine serosal surface (as above) and placental tissue seen to be invading through the surface of the uterus.

No invasion into any other organ, including the posterior wall of the bladder (a clear surgical plan can be identified between bladder and uterus).

Histologic criteria Hysterectomy specimen showing villous tissue within or breaching the uterine serosa.

Exclusion Criteria:

1. Pregnant female age more than 35 Years.
2. History of more than 3 caesarean deliveries.
3. Patient refusing conservative management.
4. Uncontrolled maternal diabetes, hypertension, Preeclampsia and Decompensated Rheumatic Heart Disease.
5. Placenta accrete( FiGO 2019 ) 8classification Grade I:

Abnormally adherent placenta (placenta adherenta or accreta) Clinical criteria Macroscopically, the uterus shows no obvious distension over the placental bed (placental "bulge"), no placental tissue is seen invading through the surface of the uterus, and there is no or minimal neovascularity Histologic criteria Microscopic examination of the placental bed samples from hysterectomy specimen shows extended areas of absent decidua between villous tissue and myometrium with placental villi attached directly to the superficial myometrium The diagnosis cannot be made on just delivered placental tissue nor on random biopsies of the placental bed.

3. Grade III(FIGO 2019)8: Abnormally invasive placenta (Percreta) Grade 3b: With urinary bladder invasion Clinical criteria At laparotomy Placental villi are seen to be invading into the bladder but no other organs. Clear surgical plan cannot be identified between the bladder a uterus. Histologic criteria Hysterectomy specimen showing villous tissue breaching the uterine serosa and invading the bladder wall tissue or urothelium.

Grade 3c: With invasion of other pelvic tissue/organ Clinical criteria At laparotomy Placental villi are seen to be invading into the broad ligament, vaginal wall, pelvic sidewall or any other pelvic organ (with or without invasion of the bladder).

Histologic criteria Hysterectomy specimen showing villous tissue breaching the uterine serosa and invading pelvic tissues/organs (with or without invasion of the bladder) For the purposes of this classification, "uterus" includes the uterine body and uterine cervix.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Estimation of blood loss | During surgery from the start of uterine incision till closure of abdominal wall
  The sum of a) Difference in Towels weighting dry & soaked . b) Volume of blood in suction apparatus. estimating the difference in Hemoglobin and Hematocrit before and after operation. estimating the number of packed red blood cells units transfused.

SECONDARY OUTCOMES:
Complication rates, | from the induction of anesthesia till 24 hours after the end of surgery
  the incidence of anesthetic, urologic injury, vascular injury, need of hysterectomy and intensive care unit admission.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sawada M, Matsuzaki S, Mimura K, Kumasawa K, Endo M, Kimura T. Successful conservative management of placenta percreta: Investigation by serial magnetic resonance imaging of the clinical course and a literature review. J Obstet Gynaecol Res. 2016 Dec;42(12):1858-1863. doi: 10.1111/jog.13121. Epub 2016 Aug 16. PMID 27527121
- [Background] Hecht JL, Baergen R, Ernst LM, Katzman PJ, Jacques SM, Jauniaux E, Khong TY, Metlay LA, Poder L, Qureshi F, Rabban JT 3rd, Roberts DJ, Shainker S, Heller DS. Classification and reporting guidelines for the pathology diagnosis of placenta accreta spectrum (PAS) disorders: recommendations from an expert panel. Mod Pathol. 2020 Dec;33(12):2382-2396. doi: 10.1038/s41379-020-0569-1. Epub 2020 May 15. PMID 32415266
- [Background] Jauniaux E, Ayres-de-Campos D, Langhoff-Roos J, Fox KA, Collins S; FIGO Placenta Accreta Diagnosis and Management Expert Consensus Panel. FIGO classification for the clinical diagnosis of placenta accreta spectrum disorders. Int J Gynaecol Obstet. 2019 Jul;146(1):20-24. doi: 10.1002/ijgo.12761. PMID 31173360